CLINICAL TRIAL: NCT06227767
Title: Investigation of the Effect of Different Intensity Stabilization Exercises on Core Muscle Stiffness and Pain in Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial
Brief Title: Investigation of the Effect of Different Intensity Stabilization Exercises on Core Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, abuzer akbaş, physiotherapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HasanKU_akbasa_001
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; core stability; ultrasonography; disability; elasticity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: two groups of exercise and a control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- exercise group twice a week (Active Comparator): Spinal stabilization exercises determined by the authors will be applied 2 days a week for 40 minutes.
  Interventions: Other: spinal stabilization exercise
- exercise group four times a week (Active Comparator): Spinal stabilization exercises determined by the authors will be applied 4 days a week for 40 minutes.
  Interventions: Other: spinal stabilization exercise
- control group (No Intervention): Patients will be followed with a home exercise program

INTERVENTIONS:
Other: spinal stabilization exercise — The exercise program will be implemented in the hospital under the supervision of a physiotherapist for 6 weeks, and the next 6 weeks will be followed as a home program. The first group will be given an exercise program 2 days a week, the second group will be given an exercise program 4 days a week. The exercise program is planned to be 40 minutes and the first 5 minutes of the program will be warm-up and the last 5 minutes will be cool-down exercises.
  Arms: exercise group four times a week; exercise group twice a week

SUMMARY:
Chronic low back pain, which individuals have difficulty coping with in the modern age and is one of the most common reasons for applying to health institutions, has important consequences for individuals and society. Approximately 80% of individuals experience low back pain throughout their lives, and 10-20% become chronic. Low back pain causes varying degrees of restrictions in individuals' daily living activities, modification or reduction of movements due to pain. This situation causes the pain to continue and causes the functional level to decrease in individuals with low back pain. There are many approaches to the treatment of chronic low back pain, and among these, exercise treatments have been shown to be effective in reducing pain and improving functionality. Spinal stabilization exercises, which have an important place among current exercise approaches for chronic low back pain, ensure the formation of a neutral position in the spine by activating the core muscles consisting of multifidus, transversus abdominis, diaphragm and pelvic floor muscles. Perception of neutral position is provided and applied in daily living activities. In this way, pain is reduced and functionality increases by providing appropriate loading. What kind of changes occur in the core muscles due to the strengthening of the core muscles as a result of spinal stabilization exercises is an important question that needs to be clarified scientifically. It is possible to observe the mechanical changes occurring in the core muscles with shear wave elastography, which has been frequently used in clinical research and practice in recent years. However, in the detailed literature review, no scientific studies were found that evaluated what level of exercise intensity produces optimal changes in the muscle and the correlation of these changes with pain and functional improvement. In this study, where different intensities of exercise will be applied, the mechanical changes occurring in the core muscles before and after exercise will be evaluated with shear wave elastography and the aim is to evaluate the correlation of these changes with pain and pain

DETAILED DESCRIPTION:
Patients with chronic low back pain who voluntarily participate in the study will be randomly divided into three groups. Physical and demographic information of the patients participating in the study will be collected. The number of patients who will participate in the study will be determined by the power analysis to be performed at the beginning of the study. Low back pain, disability index and pain sensitivity will be measured before treatment, after treatment and at the 12th week. Evaluation of core muscles with shear wave would be done at the beginning of treatment and at the 12th week. The exercise program will be implemented in the hospital under the supervision of a physiotherapist for 6 weeks, and the next 6 weeks will be followed as a home program. Participants in the first group will be included in the exercise program planned in detail below, 2 days a week, and those in the second group 4 days a week. Patients included in the third group will be followed with a home exercise program. The exercise program is planned to be 40 minutes and the first 5 minutes of the program will be warm-up and the last 5 minutes will be cool-down exercises.

In the first phase of the exercise program, patients will be placed in the hook position and contraction of the transversus abdominis muscle and multifidus muscle will be taught. Then, patients will be asked to perform exercises that enable the activation of other muscles of the body while maintaining the contraction of the transversus abdominis and multifidus muscles, and these exercises will be progressed from easy to difficult exercises. During exercise, the activation of the patients' spinal stabilizer muscles will be kept under constant control and necessary warnings will be made in this regard. Exercises will initially start with 8-10 repetitions and gradually increase to 20 repetitions. All exercises will be performed in 2 sets and there will be 30 seconds of rest between sets.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for at least 3 months.
* Not having participated in any physiotherapy or exercise program in the last month.
* Patients with informed consent

Exclusion Criteria:

* Malignancy
* Severe osteoporosis
* Arthritis
* Bone diseases
* Pregnancy
* Diabetics
* Lumbar or lower limb surgery
* Rheumatological and inflammatory problems.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of muscle elasticity with elastography | before treatment and 12nd (end of treatment) week of treatment
  The mechanical properties of the transversus abdominis, one of the core muscles, will be evaluated by the shear wave elastography method.

SECONDARY OUTCOMES:
visual analog scale | before treatment, 6th week of treatment and 12nd (end of treatment) week of treatment
  The patients' low back pain severity will be evaluated with a visual analog scale. Visual Analogue Scale: The left end of a 10 cm straight line represents no pain, and the right end represents unbearable pain. The patient will be asked to mark the pain that feels on the Visual Analog Scale ruler during the test, and then this value will be measured and recorded with the help of a ruler
oswestry disability index | before treatment, 6th week of treatment and 12nd (end of treatment) week of treatment
  In the survey, 10 pain questions evaluate the severity of pain personally, care, lifting, walking, sitting, standing, sleep, sexual life, social life, travel and the degree of change in pain. Scoring is between 0-5 for each item and items that are not answered will be excluded from evaluation.
evaluation of pain sensitivity | before treatment, 6th week of treatment and 12nd (end of treatment) week of treatment
  A pressure pain meter device (JTECH CommanderTM) will be used to evaluate pain sensitivity in patients with chronic low back pain. The measurement will be made at 3 points and the points will be 2.5 cm apart vertically on the right and left lumbar paraspinal muscles.

CONTACTS AND LOCATIONS:
Overall Officials: abuzer akbas, Principal Investigator — hasan kalyoncu university faculty of health science
Locations (2):
- Turkey (Türkiye) (2):
  - Hasan Kalyoncu University, Gaziantep, Gaziantep
  - Adıyaman training and research hospital, Adıyaman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akbas E, Ozdemir M, Akbas A, Usgu S, Bulut HT. Investigation of the effect of different intensity stabilization exercises on core muscle stiffness and pain in chronic low back pain: a single-blind, randomized controlled trial. Rheumatol Int. 2025 Aug 19;45(9):201. doi: 10.1007/s00296-025-05964-7. PMID 40828397